CLINICAL TRIAL: NCT00003078
Title: A Randomized Comparison of Radiation vs Radiation Plus Weekly Cisplatin vs Radiation Plus PVI (Protracted Venous Infusion) 5-FU in Patients With Stage II-B, III-B, and IV-A Carcinoma of the Cervix With Negative Paraaortic Nodes
Brief Title: Radiation Therapy With or Without Cisplatin or Fluorouracil in Treating Patients With Cancer of the Cervix
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065771; GOG-0165
Record Dates: First submitted 1999-11-01; First posted 2004-06-23 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2011-04

CONDITIONS: Cervical Cancer
Keywords: stage III cervical cancer; stage IIB cervical cancer; stage IVA cervical cancer; cervical squamous cell carcinoma; cervical adenocarcinoma; cervical adenosquamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Fluorouracil; Brachytherapy; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy and chemotherapy may kill more tumor cells. It is not known whether receiving radiation therapy plus cisplatin is more effective than receiving radiation therapy plus fluorouracil in treating patients with cancer of the cervix.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy plus cisplatin or fluorouracil in treating patients with primary stage IIB, stage IIIB, or stage IVA cancer of the cervix.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the progression-free survival and survival of patients with advanced cervical cancer limited to the pelvis receiving either radiotherapy alone, or radiotherapy plus weekly cisplatin, or radiotherapy plus prolonged venous infusion (PVI) of fluorouracil. [Radiotherapy alone regimen closed 8/18/98] II. Determine the relative toxic effects of radiation therapy plus chemotherapy with either weekly cisplatin or PVI fluorouracil compared to radiation alone. [Radiotherapy alone regimen closed 8/18/98] IV. Compare the progression-free survival and survival of patients with advanced cervical cancer limited to the pelvis and who smoke at the time of diagnosis versus non-smokers and those who smoke during radiation therapy versus those who quit.

OUTLINE: This is a randomized study. Patients are stratified by stage, performance of para-aortic lymphadenectomy, and brachytherapy method (HDR vs LDR). Prior to treatment patients complete a questionnaire regarding past and present smoking history and exposure to secondhand smoke. In arm I, patients undergo external radiation therapy to the pelvis once daily 5 times a week for 5 weeks. Then, patients receive either low dose rate or high dose rate intracavitary brachytherapy in one or two applications or 5 fractions once or twice a week, respectively. If intracavitary radiation therapy cannot be performed, then shrinking field technique is executed. In addition, patients receive parametrial boost once daily for 3 to 5 days during intracavitary brachytherapy. Concurrently, patients receive IV cisplatin once a week for 5 weeks beginning on day 1 of external radiation therapy and once during the parametrial boost. Patients in arm II receive external radiation therapy and brachytherapy as previously described. [Arm II closed 8/18/98] In arm III, patients undergo external radiation therapy as described in arm I. In addition, patients receive prolonged venous infusion (PVI) fluorouracil daily for 5 days during external beam radiation therapy (whole pelvis and parametrial boost). If all 6 courses of cisplatin or fluorouracil cannot be administered during external radiation therapy, then the sixth course of chemotherapy will be given during brachytherapy. Patients are followed every 3 months for the first 2 years, then every 6 months for the next 3 years, then annually until death.

PROJECTED ACCRUAL: This study will accrue a maximum of 870 patients over 66 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Primary, previously untreated, histologically confirmed invasive squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the uterine cervix stage IIB, IIIB, or IVA Negative para-aortic lymph nodes determined by lymphangiogram, CT, MRI, or lymphadenectomy (excluding suspicious para-aortic lymph nodes) Para-aortic lymphadenectomy must be performed extraperitoneally or by laparoscopy No histologically confirmed cancer involving the para-aortic lymph nodes, intraperitoneal disease, or positive peritoneal cytology No recurrent invasive carcinoma of the uterine cervix, regardless of previous treatment or cervix cancers other than squamous cell, adenosquamous, or adenocarcinoma No carcinoma of the cervical stump

PATIENT CHARACTERISTICS: Age: Any age Performance status: GOG 0-3 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times normal SGOT and alkaline phosphatase no greater than 3 times normal Renal: Creatinine no greater than 2.0 mg/dL Other: No septicemia or severe infection Not pregnant Negative pregnancy test Effective contraception required of fertile patients No other invasive malignancy unless disease free for at least 5 years and no prior cancer treatment that contraindicated this protocol therapy No concomitant malignancy other than nonmelanomatous skin cancer Must complete smoking history questionnaire and provide urine specimen for cotinine analysis

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior cytotoxic chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiation therapy to the pelvis Surgery: No prior hysterectomy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 870 (Estimated)
Dates: Start 1997-10; Primary Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachelle M. Lanciano, MD, Study Chair — Delaware County Regional Cancer Center at Delaware County Memorial Hospital
Locations (66):
- United States (65):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Women's Cancer Center, Palo Alto, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Fred J. Woods Radiation Therapy Center/St. Joseph's Cancer Institute, Tampa, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Medicine Branch, Bethesda, Maryland
  - Radiation Oncology Branch, Bethesda, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - Sooner State, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- NCIC-Clinical Trials Group, Kingston, Ontario, Canada

REFERENCES:
- [Background] Rose PG, Ali S, Whitney CW, Lanciano R, Stehman FB. Outcome of stage IVA cervical cancer patients with disease limited to the pelvis in the era of chemoradiation: a Gynecologic Oncology Group study. Gynecol Oncol. 2011 Jun 1;121(3):542-5. doi: 10.1016/j.ygyno.2011.02.024. Epub 2011 Mar 21. PMID 21420157
- [Background] Rose PG, Ali S, Whitney CW, Lanciano R, Stehman FB. Impact of hydronephrosis on outcome of stage IIIB cervical cancer patients with disease limited to the pelvis, treated with radiation and concurrent chemotherapy: a Gynecologic Oncology Group study. Gynecol Oncol. 2010 May;117(2):270-5. doi: 10.1016/j.ygyno.2010.01.045. Epub 2010 Feb 24. PMID 20181381
- [Background] Kunos C, Tian C, Waggoner S, Rose PG, Lanciano R. Retrospective analysis of concomitant Cisplatin during radiation in patients aged 55 years or older for treatment of advanced cervical cancer: a gynecologic oncology group study. Int J Gynecol Cancer. 2009 Oct;19(7):1258-63. doi: 10.1111/IGC.0b013e3181b33ace. PMID 19823064
- [Background] Gold MA, Tian C, Whitney CW, Rose PG, Lanciano R. Surgical versus radiographic determination of para-aortic lymph node metastases before chemoradiation for locally advanced cervical carcinoma: a Gynecologic Oncology Group Study. Cancer. 2008 May 1;112(9):1954-63. doi: 10.1002/cncr.23400. PMID 18338811
- [Background] Monk BJ, Tian C, Rose PG, Lanciano R. Which clinical/pathologic factors matter in the era of chemoradiation as treatment for locally advanced cervical carcinoma? Analysis of two Gynecologic Oncology Group (GOG) trials. Gynecol Oncol. 2007 May;105(2):427-33. doi: 10.1016/j.ygyno.2006.12.027. Epub 2007 Feb 2. PMID 17275889
- [Background] Gold M, Tian C, Whitney CW, et al.: Surgical versus radiologic exclusion of para-aortic lymph node metastases relative to chemoradiation for loco-regionally advanced cervical carcinoma: a meta-analysis of Gynecologic Oncology Group (GOG) protocols 85, 120 & 165. [Abstract] Society of Gynecologic Oncologists, 2006 Annual Meeting on Women's Cancer, March 22-26, 2006, Palm Springs, CA. A-39, 2006.
- [Result] Waggoner SE, Darcy KM, Tian C, Lanciano R. Smoking behavior in women with locally advanced cervical carcinoma: a Gynecologic Oncology Group study. Am J Obstet Gynecol. 2010 Mar;202(3):283.e1-7. doi: 10.1016/j.ajog.2009.10.884. Epub 2009 Dec 30. PMID 20044066
- [Result] Waggoner SE, Darcy KM, Fuhrman B, Parham G, Lucci J 3rd, Monk BJ, Moore DH; Gynecologic Oncology Group. Association between cigarette smoking and prognosis in locally advanced cervical carcinoma treated with chemoradiation: a Gynecologic Oncology Group study. Gynecol Oncol. 2006 Dec;103(3):853-8. doi: 10.1016/j.ygyno.2006.05.017. Epub 2006 Jul 3. PMID 16815535
- [Result] Lanciano R, Calkins A, Bundy BN, Parham G, Lucci JA 3rd, Moore DH, Monk BJ, O'Connor DM. Randomized comparison of weekly cisplatin or protracted venous infusion of fluorouracil in combination with pelvic radiation in advanced cervix cancer: a gynecologic oncology group study. J Clin Oncol. 2005 Nov 20;23(33):8289-95. doi: 10.1200/JCO.2004.00.0497. Epub 2005 Oct 17. PMID 16230678
- [Result] Varia MA, Bundy BN, Deppe G, Mannel R, Averette HE, Rose PG, Connelly P. Cervical carcinoma metastatic to para-aortic nodes: extended field radiation therapy with concomitant 5-fluorouracil and cisplatin chemotherapy: a Gynecologic Oncology Group study. Int J Radiat Oncol Biol Phys. 1998 Dec 1;42(5):1015-23. doi: 10.1016/s0360-3016(98)00267-3. PMID 9869224